CLINICAL TRIAL: NCT01609673
Title: Evaluation of the Early Conversion From a Calcineurin Inhibitor-based Immunosuppressive Regimen to Everolimus in de Novo Renal Transplant Recipients, a Multicenter Experience
Brief Title: Study of Everolimus in de Novo Renal Transplant Recipients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The inclusion of proposed sample turned to be infeasible due to Ethical Non-approval of 2 research sites and another site no transplant activity since 2012.
Sponsor: Helady Pinheiro, MD, PhD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Helady Pinheiro, MD, PhD, MD, PhD, Fundação Instituto Mineiro de Estudo Pesquisa Em Nefrologi
Organization: Fundação Instituto Mineiro de Estudo Pesquisa Em Nefrologi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ABR22T
Record Dates: First submitted 2012-05-24; First posted 2012-06-01 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: End Stage Renal Failure With Renal Transplant
Keywords: Immunosuppression; Chronic Kidney Disease; Renal Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): 35 patients using Cyclosporin or Tacrolimus (C0=100-200/5-10ng/mL)+ Myfortic® 1440mg/dia + Steroids.
  Medications will be administered orally, twice a day
- Intervention (Active Comparator): 35 randomized Patients Converted to Certican® (Everolimus C0=6-10 ng/mL) + Myfortic® 1440mg/day + Steroids.
  On the day of conversion (day 1), 2 mg everolimus will be introduced in the morning and at night, as morning dose of CsA or Tac will be maintained and evening dose of CsA or Tac will be reduced by 50%.
  In two days, 2 mg everolimus will be associated with 50% of CsA or Tac original dosage, both in the morning and evening. After that, everolimus dose will be adjusted to achieve a C0 target level of 6-10 ng/mL. Once target levels of everolimus are met, the CNI drug will be suspended.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — On the day of conversion (day 1), 2 mg everolimus will be introduced in the morning and at night, as morning dose of CsA or Tac will be maintained and evening dose of CsA or Tac will be reduced by 50%.
  In two days, 2 mg everolimus will be associated with 50% of CsA or Tac original dosage, both in the morning and evening. After that, everolimus dose will be adjusted to achieve a C0 target level of 6-10 ng/mL. Once target levels of everolimus are met, the CNI drug will be suspended.
  Other Names: Certican
  Arms: Intervention

SUMMARY:
In the present study, the investigators propose a conversion scheme with 50% reduction in CNI dosage until adjustment of everolimus dosage, in order to reach a trough blood level of 6-10 ng/mL, thus avoiding overimmunosuppression or alternatively breakthrough rejection episodes.

The hypothesis of this study is to demonstrate that the therapeutic regimen with Myfortic® and Certican® significantly improves renal function compared with the standard regimen of CNI.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patients
* Age between 18 and 85 years
* Recipients of living or deceased donors
* Donor under the age of 85 years
* Panel Reactivity Antibodies (PRA) over or equal to 30%
* 4-5 months post-transplant
* CNI-based immunosuppressive regimen
* Stable graft function (creatinine lower than 2.0 mg/dl)
* No currently acute rejection
* Proteinuria lower than 800mg/d
* No laboratory or physical clinically significant signs presented for the last 2 months before screening.

Exclusion Criteria:

* Recipient of multiple organs
* Recipient with a history of focal segmental glomerulosclerosis or membranous glomerulonephritis
* Presence of uncontrolled hypercholesterolemia (≥350 mg/dL)hypertriglyceridemia (over or equal to 500 mg/dL)
* Patients with eGFR lower than 40 ml/min/1.73m2
* Evidence of acute rejection within 2 months before screening
* Thrombocytopenia (lower than 75,000/mm3)
* Neutropenia (lower than 1,500/mm3)
* Leukocytopenia (lower than 2500/mm3)
* Anemia (hemoglobin lower than 6.0g/dL)
* Severe liver disease (including transaminases or bilirubin equal or over 3 times normal)
* Proteinuria over 800mg/dL
* Systemic infection or pneumonia (active infection)
* Positive for Hepatitis B, Hepatitis C or HIV.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) | 4-5 months after transplantation (baseline), and then 6 and 12 months after conversion to everolimus
  The eGFR will be calculated by Cockcroft-Gault, CKD-EPI and MDRD equations, firstly 4-5 months after transplantation (baseline), and then 6 and 12 months after conversion to everolimus (Certican ®) and suspension of CNI, associated with Myfortic ® (mycophenolate sodium enteric-coated - MSEC).

SECONDARY OUTCOMES:
graft acute rejection | 6 and 12 months after conversion
  incidence of acute biopsy-proven rejection and clinical acute rejection (without biopsy), graft loss, death with a functioning graft, and loss of follow up at 6 and 12 months after conversion;
Laboratory results and clinical alterations | 3, 6 and 12 months after conversion
  analyzing the incidence of anemia, thrombocytopenia, leukopenia, gastrointestinal side effects, pneumonitis, oral ulcers, edema, proteinuria, and any other adverse events, as well as the need of drug withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Hélady S Pinheiro, MD, PhD, Principal Investigator — Fundação IMEPEN
Locations (4):
- Brazil (4):
  - Hospital São João de Deus/Fundação Geraldo Corrêa, Divinópolis, Minas Gerais
  - Hospital Márcio Cunha/Fundação São Francisco Xavier, Ipatinga, Minas Gerais
  - Fundação IMEPEN, Juiz de Fora, Minas Gerais
  - Hospital do Rim de MOntes Claros/Irmandade Nossa Senhora das Mercês, Montes Claros, Minas Gerais